CLINICAL TRIAL: NCT00614198
Title: The ScanBrit Randomised Controlled Study of Gluten- and Casein-free Dietary Intervention for Children With Autism Spectrum Disorders
Brief Title: ScanBrit Dietary Intervention in Autism
Acronym: ScanBrit
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Center for Autisme, Denmark (Other)
Collaborators: Norway: Bo Nils og Seim Family Settlement (Unknown); The Robert Luff Foundation, United Kingdom (Unknown); Eric Birger Christensen Fond, Denmark (Unknown); Norsk Proteinintolerance, Norway (Unknown)
Responsible Party: Director Demetrious Haracopos, Center for Autisme
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA 0503g
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Results first posted 2010-10-01 (Estimated); Last update posted 2010-10-01 (Estimated); Status verified 2010-05

CONDITIONS: Autism; Autism Spectrum Disorder (ASD)
Keywords: autism; autism spectrum disorder; diet; gluten; casein; intervention; peptide; randomised; controlled; adaptive design; Autism Diagnostic Observation Schedule (ADOS); Gilliam Autism Rating Scale (GARS); Vineland Adaptive Behaviour Scale (VABS); Attention-Deficit Hyperactivity Disorder (ADHD)-IV Scale
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder; Attention Deficit Disorder with Hyperactivity | interventions — Glutens; Diet, Gluten-Free; Diet

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gluten- and casein-free diet (Experimental): Stage 1: Gluten- and casein-free dietary intervention for first 8 or 12 months. 8 or 12 months: Interim analysis based on surpassing statistical thresholds. If showed group significant improvements then progressed to stage 2 (continued on a gluten- and casein-free diet for a further 12 months).
  Interventions: Other: Gluten- and casein-free diet
- No dietary intervention (No Intervention): Stage 1: No special dietary intervention for first 8 or 12 months. 8 or 12 months: Interim analysis based on surpassing statistical thresholds. If gluten- and casein-free dietary group showed group significant improvements then progressed to stage 2 (introduction of a gluten- and casein-free diet for 12 months).

INTERVENTIONS:
Other: Gluten- and casein-free diet — Removal of foods containing gluten (cereal produce) and casein (dairy produce)
  Other Names: Gluten-free (wheat-free), casein- free (milk-free) diets
  Arms: Gluten- and casein-free diet

SUMMARY:
A growing body of research indicates that dietary intervention excluding foods containing the proteins, gluten and casein, from the diet of children diagnosed with an autism spectrum disorder (ASD) may have a positive effect on behaviour and developmental outcome.

In this single-blind, randomised-controlled, matched-pair adaptive trial, we introduced a gluten- and casein-free (GFCF) diet to a group of pre-pubescent children diagnosed with ASD concurrently with an abnormal urinary profile. Following random allocation to a diet or non- diet group, stage 1 of the study saw an intervention group follow the GFCF diet for eight months initially - progressing to 12 months if required. A non-diet control group continued with a normal diet.

Assuming significant changes for the dietary group on the various outcome measures of behaviour and development, stage 2 of the study saw both groups assigned to GFCF dietary intervention for a further 12 months when outcome measures were again assessed at study end.

DETAILED DESCRIPTION:
Eligibility criteria: diagnosis of autism, no co-morbid diagnosis of Fragile X syndrome, epilepsy or tuberous sclerosis, aged between 4-10y11m.

Experimental hypothesis: children with an autism spectrum disorder (ASD) on a GFCF diet would show a significantly improved group developmental outcome in the medium- and long-term with regards to core autism and/or secondary symptoms.

Main outcome measures: change in scores of dietary participants on one or more measures against predefined statistical thresholds as evidence of improvement, alongside changes to intra- and inter-group scores at study endpoint.

Main outcome measures ascertained by: Autism Diagnostic Observation Schedule (ADOS), Gillam Autism Rating Scale (GARS), Vineland Adaptive Behaviour Scales (VABS), Attention Deficit Hyperactivity Disorder - IV (ADHD-IV) scales.

ELIGIBILITY:
Inclusion Criteria:

* Autism Spectrum Disorder (ASD)
* Diagnosis received at Centre for Autism or a psychiatric clinic
* Abnormal urinary peptide profile

Exclusion Criteria:

* Medical treatment
* Epilepsy

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2006-04; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

REFERENCES:
- [Result] Whiteley P, Haracopos D, Knivsberg AM, Reichelt KL, Parlar S, Jacobsen J, Seim A, Pedersen L, Schondel M, Shattock P. The ScanBrit randomised, controlled, single-blind study of a gluten- and casein-free dietary intervention for children with autism spectrum disorders. Nutr Neurosci. 2010 Apr;13(2):87-100. doi: 10.1179/147683010X12611460763922. PMID 20406576
- See also: Center for Autisme, Denmark — http://www.centerforautisme.dk
- See also: ESPA Research, UK — http://www.espa-research.org.uk

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment via multiple associations
Pre-assignment Details: 92 participants were initially identified for possible study recruitment. 82 participants were available for possible study allocation; 10 participants dropped out prior to randomisation for various reasons, leaving 72 participants.
Groups:
- Gluten- and Casein-free Dietary Intervention: Stage 1: Gluten- and casein-free dietary intervention for first 8 or 12 months. 8 or 12 months: Interim analysis based on surpassing statistical thresholds. If showed group significant improvement progressed to stage 2 (continued on a gluten- and casein-free diet for a further 12 months).
- No Gluten- and Casein-free Dietary Intervention: Stage 1: No special dietary intervention for first 8 or 12 months. 8 or 12 months: Interim analysis based on surpassing statistical thresholds. If dietary intervention group showed group significant improvement progressed to stage 2 (introduction of a gluten- and casein-free diet for 12 months).
Period: Stage 1
Arm/Group | Gluten- and Casein-free Dietary Intervention | No Gluten- and Casein-free Dietary Intervention
Started | 38 | 34
Completed | 26 | 29
Not Completed | 12 | 5
Period: Stage 2
Arm/Group | Gluten- and Casein-free Dietary Intervention | No Gluten- and Casein-free Dietary Intervention
Started | 26 | 29 (Reallocated to gluten- and casein-free dietary intervention)
Completed | 18 | 17
Not Completed | 8 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gluten- and Casein-free Dietary Intervention | No Gluten- and Casein-free Dietary Intervention | Total
Number analyzed (Participants) | 38 | 34 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 38 | 34 | 72
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 8.22 (1.99) | 8.13 (2.03) | 8.15 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 33 | 31 | 64
Region of Enrollment [Number; unit: participants]
  Denmark | 38 | 34 | 72

OUTCOME MEASURES:

1. Primary Outcome: Change in Diet Groups Scores on One of Several Measures Used Against Pre-defined Statistical Thresholds as Evidence of Improvement.
Description: ADOS (Autism Diagnostic Observation Schedule): module 1 cutoff scores (communication+social): autism=12, autism spectrum (AS)=7; module 2 cutoffs: autism=12, AS=8; module 3 cutoffs: autism=10; AS=7. GARS (Gilliam Autism Rating Scale): <80 low probability of autism, 81-90 below average, 91-110 average, >110 above average probability of autism. VABS (Vineland Adaptive Behaviour Scale): <69 (low ability), 70-84 (moderate/low), 85-115 (adequate), 116-130 (moderate/high), >130 (high). ADHD-IV: 0=no problems indicated. >11 attention & >11 hyperactivity = ADHD diagnosis.
Time Frame: Baseline - 8 months - 12 months - 24 months
Population: Per protocol analysis. Analysis was conducted on n=26 (Gluten- and casein-free dietary intervention) and n=29 (No gluten- and casein-free dietary intervention) at 12 months. Analysis was conducted on n=18 and n=17 at 24 months (both on gluten- and casein-free dietary intervention).
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Gluten- and Casein-free Dietary Intervention | No Gluten- and Casein-free Dietary Intervention
Number analyzed (Participants) | 26 | 29
Units on a scale
  ADOS - Communication (8 months) | -0.16715 (0.10127) | 0.08235 (0.12096)
  ADOS - Communication (24 months) | -0.16176 (0.1204) | 0.18529 (0.11926)
  ADOS - Social (8 months) | 0.016807 (0.1024) | 0.02521 (0.12203)
  ADOS - Social (24 months) | -0.5042 (0.09795) | 0.02521 (0.13709)
  ADOS - Repetitive behaviours (8 months) | -0.14706 (0.0894) | 0.03431 (0.1139)
  ADOS - Reptitive behaviours (24 months) | -0.14216 (0.0782) | -0.0049 (0.10042)
  GARS - Social (8 months) | -1.07692 (0.29382) | -0.06897 (0.27152)
  GARS - Social (12 months) | -1.57692 (0.3097) | -0.42308 (0.36867)
  GARS - Social (24 months) | -1.88235 (0.57447) | -1.11765 (0.50645)
  GARS - Communication (8 months) | -1.23077 (0.38554) | -0.51724 (0.40203)
  GARS - Communication (12 months) | -1.47826 (0.37125) | -1.46154 (0.40089)
  GARS - Communication (24 months) | -2 (0.42875) | -1.29412 (0.60491)
  GARS - Stereotyped behaviours (8 months) | -0.96154 (0.32572) | -0.7931 (0.41338)
  GARS - Stereotyped behaviours (12 months) | -1.46154 (0.33389) | -1.3333 (0.39943)
  GARS - Stereotyped behaviours (24 months) | -0.88235 (0.44459) | -1.70588 (0.52696)
  VABS - Communication (8 months) | 0.23077 (1.35227) | 1.25 (1.73176)
  VABS - Communication (12 months) | 0.92308 (2.71629) | 1.85714 (2.05204)
  VABS - Communication (24 months) | 1.27778 (3.61895) | -2.05882 (3.19175)
  VABS - Social (8 months) | 1.53846 (2.03676) | 0.92857 (2.63369)
  VABS - Social (12 months) | -4.15385 (2.39467) | -3.25 (2.59406)
  VABS - Social (24 months) | 0.72222 (3.17033) | -3.29412 (4.29412)
  VABS - Daily Living (8 months) | 3.03846 (2.54043) | -1.64286 (2.90785)
  VABS - Daily Living (12 months) | 3.46154 (2.79903) | -2.85714 (2.8857)
  VABS - Daily Living (24 months) | -0.16667 (2.94974) | -4.64706 (4.46715)
  ADHD-IV - Inattention (8 months) | -2.15385 (0.916) | 0.31034 (0.65296)
  ADHD-IV - Inattention (12 months) | -2.19231 (0.88582) | -0.03704 (0.69488)
  ADHD-IV - Inattention (24 months) | -2.29412 (0.89016) | -3.35294 (1.14706)
  ADHD-IV - Hyperactivity (8 months) | -2.03846 (0.80667) | -0.17241 (0.60186)
  ADHD-IV - Hyperactivity (12 months) | -1.69231 (0.86606) | -0.92593 (0.55451)
  ADHD-IV Hyperactivity (24 months) | -2.58824 (1.12805) | -4.17647 (1.22845)
Statistical Analysis 1: Comparison: Gluten- and Casein-free Dietary Intervention vs No Gluten- and Casein-free Dietary Intervention; 1st stage analysis (baseline-8m or 12m) used a repeated measures model for all assessment measures. Model included baseline, age, time and time*treatment interaction. Results informed 2nd stage (8 or 12 months - 20 or 24 months). 2nd stage analysis based on various statistical scenarios (baseline vs 12 months on intervention, 12 months of no intervention vs 12 on intervention, baseline vs 24 months on intervention). No ADOS assessments were used at 12 months because of risk of practice effects; Test type: Superiority or Other; p < 0.01, Mixed Models Analysis — A priori p threshold set for stage 1 (baseline - 8m; p<0.01) or (baseline - 12 months, p<0.05) in order to progress to stage 2 (8 or 12 months - 20 or 24 months)

2. Secondary Outcome: Changes to Appearance of Multiple Compounds in Urine Samples
Time Frame: Baseline - 8 months -12 months - 24 months
Reporting Status: Not Posted
Measure: Number; unit: Participants

ADVERSE EVENTS:
Time Frame: Any indications of adverse events were continually monitored throughout the study period by study nutritionist. Assessments carried out at 8, 12 and 24 months represent periods where any adverse events could be reported.
Description: All participants on dietary intervention were potentially at mild risk from the introduction of a new dietary regime (gluten- and casein-free diet). Risk would include: disruption to eating habits & behavioural problems (associated with change to routine). Data was not collected on such mild risks.
Arm/Group | Gluten- and Casein-free Dietary Intervention | No Gluten- and Casein-free Dietary Intervention
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/34
Other Adverse Events (participants affected / at risk) | 0/38 | 0/34

LIMITATIONS AND CAVEATS:
Single-blind trial, no placebo condition, analysis based on per protocol (not intention to treat), socio-economic status not recorded, independent screening for underlying somatic conditions potentially associated with results not undertaken

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes